CLINICAL TRIAL: NCT00338871
Title: Home Based Exercise Program for Brain Injury Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: alyn1CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2007-04

CONDITIONS: Brain Injury; Cerebral Palsy
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- study (Experimental): home exercise
  Interventions: Procedure: home exercise
- control (No Intervention): regular therapy

INTERVENTIONS:
Procedure: home exercise
  Arms: study

SUMMARY:
The purpose of this study is to examine whether simple home-base aerobic exercise program have beneficial effect on walking abilities and balance performance in children with brain damage

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of CP or ABI Must be able to stand with or without aid.

Exclusion Criteria:

Can not follow simple commands

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Katz-Leurer, PhD, Study Director — Alyn Hospital Jerusalem
Locations (1):
- Alyn Pediatric and Adolesencent Rehabilitation Center, Jerusalem, Israel